CLINICAL TRIAL: NCT03942185
Title: Chinese Herbal Medicine for the Treatment of Psoriasis Vulgaris: a Real World Study
Brief Title: Chinese Herbal Medicine for Psoriasis Vulgaris: a Real World Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Zhejiang Provincial Hospital of TCM (Other); Shanghai Dermatology Hospital (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Changhai Hospital (Other); Shanghai 10th People's Hospital (Other); Beijing Hospital of Traditional Chinese Medicine (Other); Wuhan No.1 Hospital (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Chinese Medicine Hospital Affiliated to Southwest Medical University (Unknown); First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other); The Second Affiliated Hospital of Jiangxi University of TCM (Unknown); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); The Guangxi Zhuang Autonomous Region Institute of Dermatology and control (Unknown); The First Affiliated Hospital of Guiyang College of TCM (Unknown); The Second People's Hospital Affiliated to Fujian University of TCM (Unknown); Gansu University of Chinese Medicine (Other); Shanxi Provincial Hospital of Traditional Chinese Medicine (Unknown); Shijiazhuang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018YFC1705301
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Psoriasis
Keywords: Psoriasis Vulgaris; Chinese Medicine; Real World Study; Clearing heat and Cooling blood; Promoting blood circulation and Removing blood stasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Psoriasis with Blood heat syndrome group (Experimental): Participants in Psoriasis with Blood heat syndrome group will receive Chinese Herbal Medicine internal treatment according with the Chinese Medicine principle of Clearing heat and Cooling blood, such as Cool blood detoxification Decoction I，Cool blood and activating blood prescription compound, Cool blood detoxification Decoction II, Cool blood activating blood Decoction, Tufu drink, Xiaoyin Decoction and etc., two times per day for 8 weeks.
  Interventions: Drug: Oral Chinese Herbal Medicine of Clearing heat and Cooling blood therapy
- Psoriasis with Blood stasis syndrome group (Experimental): Participants in Psoriasis with Blood stasis syndrome group will receive Chinese Herbal Medicine internal treatment according with the Chinese Medicine principle of Promoting blood circulation and Removing blood stasis, such as Huoxue Sanyu Xiaoyin Decoction, Cool blood detoxification Decoction III and etc., two times per day for 8 weeks.
  Interventions: Drug: Oral Chinese Herbal Medicine of Promoting blood circulation and Removing blood stasis therapy
- Psoriasis with Non-Blood heat or Blood stasis syndrome group (Experimental): Participants in Psoriasis with Non-Blood heat or Blood stasis syndrome group will receive Chinese Herbal Medicine internal treatment according with the Chinese Medicine principle of syndrome differentiation therapy two times per day for 8 weeks.
  Interventions: Drug: Oral Chinese Herbal Medicine according with syndrome differentiation therapy
- Healthy control group (No Intervention): No Intervention.

INTERVENTIONS:
Drug: Oral Chinese Herbal Medicine of Clearing heat and Cooling blood therapy — Oral Chinese Herbal Medicine of Clearing heat and Cooling blood therapy, warm water decoction, 1 dose/day, divided into 2 times, 180 ~ 200ml each time for 8 weeks.
  Arms: Psoriasis with Blood heat syndrome group
Drug: Oral Chinese Herbal Medicine according with syndrome differentiation therapy — Oral Chinese Herbal Medicine according with syndrome differentiation therapy, warm water decoction, 1 dose/day, divided into 2 times, 180 ~ 200ml each time for 8 weeks.
  Arms: Psoriasis with Non-Blood heat or Blood stasis syndrome group
Drug: Oral Chinese Herbal Medicine of Promoting blood circulation and Removing blood stasis therapy — Oral Chinese Herbal Medicine of Promoting blood circulation and Removing blood stasis therapy, warm water decoction, 1 dose/day, divided into 2 times, 180 ~ 200ml each time for 8 weeks.
  Arms: Psoriasis with Blood stasis syndrome group

SUMMARY:
The purpose of this study is to establish a multi-center clinical registration platform, to form the real world evidence of New Blood Syndrome Theory intervention in psoriasis, and to evaluate the therapeutic advantages of New Blood Syndrome Theory therapy in the clinical effective and recurrence rate of psoriasis vulgaris.

DETAILED DESCRIPTION:
Psoriasis is a common chronic and recurrent inflammatory skin disease. The incidence of the disease is increasing year by year, seriously affecting people's quality of life. The systematic treatment of psoriasis in modern medicine is limited of wide application due to the adverse reactions of different degrees and the high economic cost.

Chinese Medicine (CM) has unique advantages in treatment of psoriasis. On the basis of CM principle--"Blood Differentiation and Treatment" in psoriasis and the combination of clinical experience, Chinese famous professor Wanzhang Qin proposed the "New Blood Syndrome Theory" in psoriasis--the psoriasis based in blood, with blood heat first, and blood stasis throughout the whole process of psoriasis. This study will form a systematic report on the diagnosis and treatment of psoriasis with the New Blood Syndrome Theory; theoretically verified by prospective cohort studies, a theoretical system of the New Blood Syndrome Theory for psoriasis will be constructed.

Objectives of this study are to establish a multi-center clinical registration platform, to form the real world evidence of New Blood Syndrome Theory intervention in psoriasis, and to evaluate the therapeutic advantages of New Blood Syndrome Theory therapy in the clinical effective and recurrence rate of psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria of psoriatic:

1. In line with the western and Chinese Medicine diagnosis standard of psoriasis vulgaris and Chinese Medicine syndrome diagnosis standard of psoriasis;
2. 18 to 65 years old, male or female patient;
3. The selected subjects cannot be selected or omitted until the pre-designed number of cases is completed;
4. Informed consent must be obtained.

Exclusion Criteria of psoriatic:

1. Patients with a history of serious mental illness or family history;
2. Other reasons that the investigator considered inappropriate to participate in the study.

Inclusion Criteria of health volunteers:

1. Not in line with the western and Chinese Medicine diagnosis standard of psoriasis vulgaris and Chinese Medicine syndrome diagnosis standard of psoriasis;
2. 18 to 65 years old, male or female patient;
3. The selected subjects cannot be selected or omitted until the pre-designed number of cases is completed;
4. Informed consent must be obtained.

Exclusion Criteria of health volunteers:

1. Other active skin diseases which may affect the condition assessment are present;
2. Those with severe, uncontrollable local or systemic acute or chronic infections;
3. Patients with a history of serious mental illness or family history;
4. Other reasons that the investigator considered inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | Up to 56 days after treatment
  Psoriasis Area and Severity Index involves grading psoriatic plaques based on erythema (E), infiltration (I), desquamation (D). Severity is graded from 0-4 for each criteria (0 - none, 1 - slight, 2 - moderate, 3 - severe, and 4 - very severe). The body is divided into 4 regions, head, upper extremities, trunk, and lower extremities, and for each region, the surface area involvement is graded on a 0-6 scale (0 - 0% involvement, 1 - <10%, 2 - 10-<30%, 3 - 30-<50%, 4 - 50-<70%, 5 - 70-<90%, 6 - 90-100%).The highest potential PASI score is 72, with higher PASI scores indicating worse psoriasis.

SECONDARY OUTCOMES:
Body surface area (BSA) | Up to 56 days after treatment
  The percentage of BSA involved in psoriasis is estimated by fingerprinting, where the entire palm of the patient represents approximately 1% of the total BSA. The number of handprints on psoriasis skin in a body part is used to determine the extent to which the body part is affected by psoriasis (%).
Physician Global Assessment (PGA) | Up to 56 days after treatment
  Physician Global Assessment (PGA) is scored on a 5-point scale, reflecting a global consideration of the erythema (E), infiltration (I), desquamation (D) across all psoriatic lesions. It is calculated as follows: PGA score = (E + I + D) / 3, then the score needs to be rounded to the nearest whole number [PGA scale: Clear (0) - Very Severe (5)].
Dermatology Life quality index(DLQI) | Up to 56 days after treatment
  The Dermatology Life Quality Index (DLQI) is a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores range from 0-30, a higher score indicating a greater impact on a participant's quality of life.
Patient-reported quality of life (PRQoL) | Up to 56 days after treatment
  PRQoL is used to assess the impact of psoriasis on individual social life. Scores range from 0-25, a higher score indicating a greater impact on a participant's social life.
Visual Analogue Score (VAS) | Up to 56 days after treatment
  Visual Analog Scale (VAS) is used to measure lesion pruritus from 0 to 100 mm at eash visit (with 0 being no pruritis and 100 being maximum pruritis).
CM symptom score | Up to 56 days after treatment
  The CM symptom score is used to assess changes in blood syndrome related symptoms during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Chair — Department of dermatology, Shanghai Yueyang Integrated Medicine Hospital, Shanghai
Locations (20):
- China (20):
  - The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine, Hefei, Anhui
  - Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - The Second People's Hospital Affiliated to Fujian University of TCM, Fuzhou, Fujian
  - Affiliated Hospital of Gansu University of traditional Chinese Medicine, Lanzhou, Gansu
  - The Guangxi Zhuang Autonomous Region Institute of Dermatology and control, Nanning, Guangxi
  - The First Affiliated Hospital of Guiyang College of TCM, Guiyang, Guizhou
  - Shijiazhuang Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - First Affiliated Hospital of Heilongjiang Chinese Medicine University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Affiliated hospital of jiangxi university of traditional Chinese medicine, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Jiangxi University of TCM, Nanchang, Jiangxi
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Hospital of Traditional Chinese Medicine, Xi’an, Shanxi
  - Chinese Medicine Hospital Affiliated to Southwest Medical University, Luzhou, Sichuan
  - Zhejiang Provincial Hospital of TCM, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun X, Zhao H, Wang R, Li H, Wu Y, Ze K, Su Y, Li B, Li X. Psoriasis complicated with metabolic disorder is associated with traditional Chinese medicine syndrome types: a hospital-based retrospective case-control study. Curr Med Res Opin. 2023 Jan;39(1):19-25. doi: 10.1080/03007995.2022.2129803. Epub 2022 Oct 11. PMID 36189747
- [Derived] Luo Y, Ru Y, Sun X, Zhou Y, Yang Y, Ma T, Xu R, Chen J, Zhou M, Ze K, Ju L, Wang Y, Yin Q, Wang R, Li B, Li X. Characteristics of psoriasis vulgaris in China: a prospective cohort study protocol. Ann Transl Med. 2019 Nov;7(22):694. doi: 10.21037/atm.2019.10.46. PMID 31930095